CLINICAL TRIAL: NCT01385345
Title: Can Vitamin D Replacement Reduce Insulin Resistance In South Asians With Vitamin D Deficiency?
Brief Title: Vitamin D Replacement in Insulin Resistant South Asians
Acronym: VITALITY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recommended by DMEC. Poor recruitment, changes in current clinical management of Vit D deficiency. Research question no longer relevant
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0166
Record Dates: First submitted 2011-06-14; First posted 2011-06-30 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2013-01

CONDITIONS: Vitamin D Deficiency; Insulin Resistance
Keywords: Vitamin D deficiency; Insulin resistance
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 high dose (Active Comparator): 200,000 units (time 0) followed by (100,000 units) at months 1.5, 3 and 5. Participants will also have daily 1,000 units per day to mirror the control arm and maintain double blinding.
  Interventions: Drug: Vitamin D3 cholecalciferol
- Vitamin D3 (Placebo Comparator): Participants will have a placebo liquid (to mirror the active arm high dose Vitamin D3) and also have daily 1,000 units Vitamin D3.
  Interventions: Drug: Vitamin D3 cholecalciferol

INTERVENTIONS:
Drug: Vitamin D3 cholecalciferol — High dose Vitamin D3 (200,000 units followed by 100,000 units x 3 over 6 months) plus daily 1,000 units Vitamin D3 per day vs only daily 1,000 units Vitamin D3 per day

SUMMARY:
This study will test the hypothesis that 6 months of periodic high dose Vitamin D3 replacement (200,000 and 100,000 units cholecalciferol, oral liquid drops at 6 to 8 week intervals) followed in-between by daily 1000 units, decreases insulin resistance by HOMA2-IR ≥ 0.36, in comparison to control, standard dose Vitamin D3 1000IU/ day for 6 months, in south Asians with both Vitamin D deficiency (defined as 25 Hydroxy vitamin D < 25nmol/l) and insulin resistance (defined as HOMA1 -IR≥ 1.93).

The hypothesis formed suggests that insulin resistance developed in South Asians is explained, at least in part, by the presence of Vitamin D Deficiency (VDD). Therefore if the VDD is reversed/ 'normalised into target range' using Vitamin D therapy in individuals at risk of diabetes, then markers of insulin resistance should reduce from baseline values. However, current UK recommended doses of Vitamin D do not adequately replenish severe VDD, common in South Asians, back into the target range and therefore will not reduce insulin resistance markers. Therefore only higher pharmacological doses are able to replace severe Vitamin D deficiency adequately and improve insulin resistance markers.

DETAILED DESCRIPTION:
Cardio metabolic risk in South Asians

Incident Cardiovascular Disease (CVD) within the South Asian Diaspora has failed to decline in parallel with other migrant groups. Rates of coronary disease in middle-aged South Asians, 50% higher than UK background, are concerning and place a growing socio-economic burden on communities and health-care providers. Concerted efforts to recognise and manage early CVD-risk within this highly susceptible group are essential if persistent health inequalities are to be adequately addressed. Significant variation in CVD implies differential interaction of risk factors across populations or the presence of additional factors accounting for increased risk. Metabolic conditions prevalent in South Asians and characterised by insulin resistance, glucose disorders and dyslipidaemia may be key to addressing observed CVD differences. Type 2 Diabetes Mellitus (T2DM) develops early in South Asians and once established carries a high risk of vascular mortality. Prediabetes is more common in South Asians and associate independently with vascular and diabetes-risk. Ethnic pre-disposition to central obesity and its metabolic consequences is clearly important in determining CVD risk, but even when combined with other factors (e.g. social-economic deprivation, smoking, blood pressure) fails to entirely account for observed variation in vascular events between groups. Assumptions that cultural incompatibility and medication compliance influence CVD outcomes are largely unsubstantiated, implying unidentified factors contribute to increased risk in South Asians.

Vitamin D Deficiency (VDD)

There has been a resurgence of interest in the recognition and treatment of VDD beyond established roles in metabolic bone disease. Epidemiological studies implicate vitamin D and calcium homeostasis in a plethora of non-skeletal immune-based chronic diseases. Proposed mechanisms accounting for these pleiotropic actions focus upon well-characterised in-vitro immuno-modulatory effects, intracellular calcium signalling and the recent finding that the Vitamin D receptor is ubiquitous. The emerging science connecting biochemical deficiency, molecular or cytokine responses and disease pathogenesis is well-reviewed. VDD appears to predispose to vascular, rheumatic and neuropathic inflammation, hypertension, metabolic syndrome and atherosclerosis.

Data from large observational cohorts and trials designed for bone-related outcomes consistently demonstrate inverse relationships between (1) serum 25-hydroxy-cholecalciferol (25(OH)VitD) and prevalent T2DM/CVD or conversely, (2) supplementation and incident all cause mortality. Baseline serum 25(OH)VitD predicts future glycaemic status, whilst VDD associates with markers of insulin resistance, coronary calcification, aortic stiffness, left ventricular mass, endothelial dysfunction, and hypertension. Diabetes-related micro and macro-vascular complications may be exacerbated by VDD.

Reported Vitamin D intervention studies have so far been limited by small sample sizes, inadequate replacement and short intervention times. Whist variability of study populations, dosage regimes and endpoints has made comparison of available intervention data difficult, for metabolic outcome trends definitely favour enhanced insulin sensitivity and action. One study using 700 IUD3 daily for two years, demonstrated glucose reduction in IFG comparable with intensive lifestyle intervention of the Diabetes Prevention Project.

Conversely the WHI study failed to demonstrate any Vitamin D effects on either glycaemic or blood pressure outcomes with a possibly sub-therapeutic 400 IU daily replacement which increased serum 25(OH)Vitamin D by an average of 7nmol/l. In the absence of well-designed supplementation trials, the strongest evidence continues to lie with prospective association studies that can neither confirm causality nor exclude confounding influences.

The optimal Vitamin D level is defined as >75nmol/l, adequate level 50-75nmol/l, sub-optimal 25-50nmol/l and deficient <25nmol/l.

The South Asian VDD phenotype

It is plausible T2DM and CVD prevalence in South Asians relates directly to sub-optimal Vitamin D status. This population is ideal for prospective phenotyping and intervention trials as it remains the largest reservoir of endemic VDD in the UK (Leicester population data: 72% 25(OH) Vitamin D < 20 nmol/l).

Recognised causes of VDD susceptibility in South Asians include 1) skin complexion, 2) lack of sunlight exposure, 3) vegetarianism, and 4) adipose tissue vitamin sequestration, although surprisingly there is lack of evidence supporting a specific dosing regime in this Vitamin D deplete population. Consensus algorithms for replacement based predominantly on bone-related outcomes in Caucasians are unlikely to adequately address VDD in South Asians, nor indeed associated cardio-metabolic effects based upon the currently available trial evidence. The prospect of vitamin D supplementation as a potential intervention for both diabetes and other cardiovascular risk factors carries considerable public health implication. Far from an ethnic minority niche, VDD prevalence is set to rise in line with Western obesity trends. It is therefore imperative the investigators determine the potential of this most simple of treatments in the prevention of cardio-metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

We will include the following people if they meet all criteria:

1. 25-75 year old south Asian (Bangladeshi, Indian or Pakistani) men or women.
2. A low vitamin D level (defined by a specific marker, 25(OH)VitD <25 nmol/L)
3. Insulin resistance, defined as homeostatic model assessment of Insulin resistance (HOMA1-IR) ≥ 1.93.

Exclusion Criteria:

We will exclude people if they have any one of the following:

1. Those who have been told by a doctor they have diabetes (Type 1 or 2).
2. Those who developed new diabetes (World Health Organisation (WHO) 1999 guidelines) detected on the Screening Visit fasting glucose test (such participants will be offered a confirmatory test to determine if they have diabetes with an oral glucose tolerance test) or the oral glucose tolerance test at Baseline Visit. Any individual with new diabetes will have follow up arranged with a doctor. If the confirmatory test does not show new diabetes, the participant will is eligible to re-enter the study.
3. HbA1c ≥ 7.0% which is suggestive of diabetes.
4. Pre-existing calcium and/or Vitamin D tablets (D2 ergocalciferol or D3 cholecalciferol) / therapy (e.g. intramuscular injections, oral liquid preparations) or previous adverse reaction to Vitamin D (D2 or D3). Any individual who has previously been on these therapy must have been off Vitamin D/ Calcium for at least six months.
5. Pregnancy or breast feeding females, or actively trying/ intending to become pregnant during the planned six month trial.
6. A history of known or newly detected hypercalcaemia or hypocalcaemia, hyperparathyroidism (that induce high calcium levels), kidney stones or other kidney problems/ low kidney function (estimated glomerular filtration rate <60 = Chronic kidney disease stage 3, 4 or 5) or known history of liver problems/ disorders.
7. A history of known bone diseases (e.g. osteoporosis, osteomalacia, osteopetrosis) or muscle diseases.
8. Any participant discovered to have new kidney/ liver/ bone or other health problems discovered during Screening or Baseline visit. Such individuals will have appropriate follow up organised. A raised Parathyroid Hormone (PTH) will be considered in the clinical context of symptoms, Alkaline Phosphatase (ALP) and Vitamin D level (i.e. may or may not be excluded).
9. Terminal illness, malignancy or physical inability to give consent (not language barriers).
10. Taking medications which may interfere with Vitamin D metabolism (phenytoin, carbamazepine, primidone and barbiturates) or potentially leading to other problems (bendroflumethiazide, digoxin).
11. Participants unable to commit time for the six month study (e.g. holiday abroad, work commitments).
12. Actively taking part in another interventional study (e.g. medication, lifestyle Randomised controlled trials); observational and cross sectional studies are still permitted.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
HOMA2-IR (homeostatic model assessment of insulin resistance) | 6 months
  This study will test the hypothesis that 6 months of periodic high dose Vitamin D3 replacement (200,000 and 100,000 units cholecalciferol, oral liquid drops at 6 to 8 week intervals) followed in-between by daily 1000 units, decreases insulin resistance by HOMA2-IR ≥ 0.36, in comparison to control, standard dose Vitamin D3 1000IU/ day for 6 months, in south Asians with both Vitamin D deficiency (defined as 25 Hydroxy vitamin D < 25nmol/l) and insulin resistance (defined as HOMA1 -IR≥ 1.93).

SECONDARY OUTCOMES:
fasting plasma glucose | 6 months
  reduction in fasting plasma
HbA1c | 6 months
two hour plasma glucose | 6 months
Tolerability of high dose Vitamin D3 treatment regime | 6 months
  We will assess how tolerable taking the high dose Vitamin D3 treatment in terms of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom